CLINICAL TRIAL: NCT06306443
Title: A Comparative Effectiveness Trial of Sublingual Versus Extended-release Buprenorphine With Individuals Leaving a Carceral Setting
Brief Title: Buprenorphine for Individuals in Jail
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20235453
Record Dates: First submitted 2024-02-28; First posted 2024-03-12 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- extended-release buprenorphine (XR-B) (Experimental): Participants will receive sublingual (sl; taken under the tongue) buprenorphine/naloxone doses of 2 mg for two days followed by 4mg for 2 days. The speed of induction will be based on their response to sl buprenorphine/naloxone. If they tolerate sl buprenorphine, on day 4 they will be administered an 8 mg dose of BRIXADI on day 5 (if they do not tolerate sl buprenorphine/naloxone we will extend sl dosing). During week two of dosing, they will receive 16 mg dose of BRIXADI will be given, based on the participant's response to the previous dose. During week three of dosing, they will receive a 24 mg dose of BRIXADI. During week four they will be administered a monthly dose of 64mg, 96mg, or 128mg. In all cases, the dose selected will be based on their response to the previous weeks' dose. We will endeavor to get you on the 96 mg or 128 mg monthly dose as there is a lack of opioid blockade data for the 64 mg monthly dose.
  Interventions: Drug: extended-release buprenorphine (XR-B)
- sublingual buprenorphine (SL-B) (Active Comparator): Participants will receive sublingual (sl; taken under the tongue) buprenorphine/naloxone doses of 2 mg for two days followed by 4mg for 2 days. The speed of induction will be based on their response to sl buprenorphine/naloxone.
  Interventions: Drug: extended-release buprenorphine (XR-B)

INTERVENTIONS:
Drug: extended-release buprenorphine (XR-B) — buprenorphine
  Other Names: sublingual buprenorphine (SL-B)

SUMMARY:
This study is an open label randomized controlled trial of extended-release buprenorphine (BRIXADI, XR-B) vs. sublingual buprenorphine (SL-B) in a large metropolitan jail. An open-label design will randomly assign 240 adults with moderate-to-severe OUDs who are soon-to-be-released from jail to either XR-B (n=120) or SL-B (n=120) treatment in jail followed by 6-months of post-release buprenorphine treatment, a 7-month safety visit, and a final long-term follow-up at 12-months.

DETAILED DESCRIPTION:
This study is an open label randomized controlled trial of extended-release buprenorphine (BRIXADI, XR-B) vs. sublingual buprenorphine (SL-B) in a large metropolitan jail. An open-label design will randomly assign 240 adults with moderate-to-severe OUDs who are soon-to-be-released from jail to either XR-B (n=120) or SL-B (n=120) treatment in jail followed by 6-months of post-release buprenorphine treatment, a 7-month safety visit, and a final long-term follow-up at 12-months.

Aim 1. Compare the effectiveness of XR-B vs. SL-B Aim 2. To calculate the cost to the state and/or jail/city health system of implementing XR-B and SL-B, and determine the relative value, including the costs associated with the interventions in the community, from a county and state-policymaker and societal perspective.

Aim 3. Explore barriers and facilitators to XR-B versus SL-B implementation in jail: (1) dose induction; (2) diversion and procedures for reducing diversion; (3) continuity of care after release or transfer to another facility; (4) staffing (both custody and medical) needs for daily versus XR-B buprenorphine dosing; and (5) patient preference for XR-B versus SL-B.

Primary Outcome. (a) illicit opioid use (i. urine toxicology; ii. self-reported days of opioid use using Timeline Followback; and iii. time to opioid relapse).

Secondary Outcomes. (b) retention in buprenorphine treatment (i. days receiving buprenorphine and ii. time to treatment dropout); (c) other illicit substance use (i. urine toxicology; ii. self-reported days of illicit substance use using Timeline Followback; (d) overdose events (non-fatal and fatal); (e) quality of life (i. physical health; ii. mental health); (f) HIV risk behaviors (i. sexual risk behavior; ii. needle use or sharing); and (g) criminal activity (i. crime days; ii. re-arrest; iii. technical violations; iv. re-incarceration).

Costs. (a) cost to the correctional system; (b) costs associated with community intervention

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female inmates at participating jail who are eligible for release within 120 days (sentenced and/or pretrial [note: individuals who might be sentenced to state/federal prison will be excluded]); Those individuals who are pre-trial and/or sentenced who are completing their sentence in the community (probation, parole, home detention, electronic monitoring, drug or other treatment court [or equivalent]) will be eligible to participate;
* History of opioid use disorder (meeting DSM-5 criteria of moderate or severe opioid use disorder at the time of incarceration; individuals not meeting the opioid-disorder criterion will be eligible if they were treated in an opioid agonist treatment program during the year before incarceration);
* Suitability for XR-B and/or SL-B treatment as determined by medical evaluation;
* Willingness to enroll in XR-B or SL-B treatment in jail and continue in the community;
* Planning to live in Baltimore City or the Baltimore Region;

Exclusion Criteria:

* Liver function test levels greater than 5 times normal (if we are unable to obtain labs, a determination by the study physician will be made to allow inclusion);
* Active medical illness that may make participation hazardous (e.g., unstable diabetes, heart disease; moderate to severe renal impairment; adequately treated medical conditions are acceptable);
* Conditions or medications that may predispose to QTc prolongation (personal or family history of long QT syndrome, hypokalemia, medications that prolong QTc interval, e.g., macrolide antibiotics, azole antifungal compounds, anti-arrythmics, antipsychotics and antidepressant);
* Untreated psychiatric disorder that may make participation hazardous (e.g., untreated psychosis, bipolar disorder with mania; adequately treated psychiatric disorders and appropriate psychotropic medications will be allowed);
* History of allergic reaction to buprenorphine;
* Suicidal ideation (within the past 6 months);
* Inability to pass a study enrollment quiz; and
* Currently receiving non-buprenorphine MOUD in jail (methadone, naltrexone).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
urine toxicology | 12-months
  positive urine drug screen for opioids
days of opioid use | 12-months
  Number of days since last assessment
time to opioid relapse | 12-months
  days from release from jail to first relapse event

SECONDARY OUTCOMES:
retention in buprenorphine treatment | 6-months
  days receiving buprenorphine
urine toxicology for other illicit substance use | 12-months
  positive urine drug screen
days of illicit substance use | 12-months
  number of days since last assessment
overdose events | 12-months
  fatal and non-fatal overdose events
PROMIS Patient-Reported Outcomes Measurement Information System - physical health | 12-months
  Global physical health score
PROMIS Patient-Reported Outcomes Measurement Information System - mental health | 12-months
  Global mental health score
HIV risk behaviors (Risk Assessment Battery, RAB) - sex risk score | 12-months
  sexual risk behavior; Scored 0-18 (higher risk)
HIV risk behaviors (Risk Assessment Battery, RAB) needle use or sharing score | 12-months
  needle use or sharing; Scored 0-22 (higher risk)
criminal activity | 12-months
  i. crime days; ii. re-arrest; iii. technical violations; iv. re-incarceration

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Friends Research Institute, Baltimore, Maryland
  - Baltimore Central Booking & Intake Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Working on a plan.